CLINICAL TRIAL: NCT02801149
Title: A Single Centre Randomised, Non-blinded, Prospective Study to Evaluate the Use of MRI for Patients Presenting With Suspected Scaphoid Fracture With Negative Findings on the Initial Conventional Radiography
Brief Title: The Use of MRI in the Assessment of Suspected Scaphoid Fracture With Negative Findings on the Initial Plain Radiography
Acronym: SMRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Scaphoid MRI
Record Dates: First submitted 2016-06-03; First posted 2016-06-15 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Scaphoid Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No further imaging (No Intervention): Patients randomised to this group will receive standard care, i.e. will not undergo additional imaging scans at A&E/Urgent Care Centre.
- Wrist Magnetic Resonance Imaging (MRI) (Experimental): Patients randomised to this group will undergo an additional 3-sequence wrist MRI during the initial A&E/Urgent Care Centre episode.
  Interventions: Procedure: Wrist Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Procedure: Wrist Magnetic Resonance Imaging (MRI) — Patients that enter this group are randomised to receive non-standard care with a 3-sequence MRI scan of the scaphoid following the initial conventional radiography.
  Arms: Wrist Magnetic Resonance Imaging (MRI)

SUMMARY:
Given that: 1) various clinical complications may arise from a misdiagnosed scaphoid fracture; and 2) clinical and radiographic diagnosis of scaphoid fracture is often challenging, particularly at the time of presentation, this study aims to evaluate whether the use of Magnetic Resonance Imaging (MRI) in the investigation of patients presenting with a suspected scaphoid fracture, with negative findings from the initial conventional radiography (4-view plain x-ray), leads to improved levels of efficiency, quality of care and patient experience.

This study is a single centre randomised, non-blinded, prospective study. Participants will be randomised, following the initial negative conventional radiography, to either: no further imaging at A&E (consistent with current clinical practice); or 2) wrist MRI. The study considers a follow-up period of 6 months.

DETAILED DESCRIPTION:
The scaphoid bone is an obliquely orientated bone on the radial (thumb) side of the wrist, between the distal carpal row and the radius. Wrist injury is a common presentation to the Emergency Department (ED) in the UK. Amongst these patients, the scaphoid is the most commonly fractured carpal bone, accounting for 51-90% of carpal fractures and between 2-7% of all fractures.

Given that: 1) various clinical complications may arise from a misdiagnosed scaphoid fracture; and 2) clinical and radiographic diagnosis of scaphoid fracture is often challenging, particularly at the time of presentation, this study aims to evaluate whether the use of Magnetic Resonance Imaging (MRI) in the investigation of patients presenting with a suspected scaphoid fracture, with negative findings from the initial conventional radiography (4-view plain x-ray), leads to improved levels of efficiency, quality of care and patient experience.

This study is a single centre randomised, non-blinded, prospective study. Participants will be randomised, following the initial negative conventional radiography, to either: no further imaging at A&E (consistent with current clinical practice); or 2) wrist MRI. The study considers a follow-up period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

Every patient aged 16 years or over presenting at A&E/UCC with clinical history and examination consistent with a suspected scaphoid fracture but negative findings on the initial 4-view plain x-ray. It is considered that a patient has suspected scaphoid fracture if at least one of the following criteria are present:

* Isolated pain / tenderness over the Anatomical Snuff Box (ASB) or Scaphoid Tubercle or pain in the scaphoid region during axial loading of the 1st metacarpal.
* History of recent fall (< 14 days) on an out-stretched hand (FOOSH), wrist injury or poor history associated with examination findings suggestive of scaphoid fracture.

Furthermore, only patients that present at A&E/UCC during the following schedule of MRI normal working hours will be included in the study:

* Patients screened for the study at A&E/UCC on weekdays after 7.30 am and before 6 pm;
* Patients screened for the study at A&E/UCC on weekends or Bank Holidays after 9 am and before 4 pm.

Exclusion Criteria:

* Patients presenting outside GSTT's catchment area who are not willing to be followed-up at GSTT;
* Patients with a confirmed scaphoid fracture following the initial 4-view plain x-ray;
* Patients with confirmed ipsilateral upper limb injury/injuries (e.g. wrist/forearm/arm injury) following initial conventional x-ray examination(s) - regardless of the findings around the suspected scaphoid fracture.
* Patients with suspected scaphoid fracture not admitted through A&E at St Thomas' Hospital or Urgent Care Centre (UCC) at Guy's Hospital;
* Patients who lack capacity to give consent or participate in the study;
* Patients that are already taking part in a Clinical Trial of an Investigational Medicinal Product (CTIMP);
* Prisoners.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2016-06-06 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
3-month costs (measured in £ per patient) associated with the two clinical groups following the A&E/UCC initial episode | 3 months
  The primary objective is to estimate the 3-month costs associated with two clinical pathways at A&E/UCC: (i) the current pathway, with x-ray as the only imaging modality (no further imaging group); or (ii) the proposed pathway (MRI group), with a hybrid approach i.e. using x-ray as the initial imaging modality and subsequently MRI for patients with negative findings on the initial x-ray.

SECONDARY OUTCOMES:
6-month costs (measured in £ per patient) associated with the two clinical groups following the A&E/UCC initial episode | 6 months
  This objective aims to estimate the 6-month costs associated with two clinical pathways at A&E/UCC: (i) the current pathway, with x-ray as the only imaging modality (no further imaging group); or (ii) the proposed pathway (MRI group), with a hybrid approach i.e. using x-ray as the initial imaging modality and subsequently MRI for patients with negative findings on the initial x-ray.
3-month cost-effectiveness analysis (ICER measured as £ per QALY) following the A&E/UCC initial episode | 3 months
  A cost-effectiveness analysis takes into account both the costs and outcomes related to the interventions. An unique incremental cost-effectiveness ratio (ICER), measured as £ per QALY, will be estimated comparing both interventions at 3 months.
6-month cost-effectiveness analysis (ICER measured as £ per QALY) following the A&E/UCC initial episode | 6 months
  A cost-effectiveness analysis takes into account both the costs and outcomes related to the interventions. An unique incremental cost-effectiveness ratio (ICER), measured as £ per QALY, will be estimated comparing both interventions at 6 months.
Cost per correctly diagnosed scaphoid fracture (measured in £ per correct diagnosis) | 3 months
  The cost per correctly diagnosed scaphoid fracture with the proposed intervention compared to standard care will be considered to evaluate whether overall potential cost-savings are aligned with the benefits of an improved diagnostic pathway.
  Findings from the treatment group (with MRI) and the control group (no further imaging) will be compared against the 3-month 4-view plain x-ray (gold standard). If both imaging findings are consistent, it is considered that a correct diagnosis was achieved.
Patient satisfaction in both groups (to be assessed using non-standard questionnaires, based on a 1-5 likert scale) | 3 months
  Patient experience will be evaluated using patient questionnaires. The underlying hypothesis is that the use of MRI will promote an improvement in the patient's overall experience, due to: i) a decrease in the need for secondary care contacts; ii) the reduction of plaster casts utilisation; and (iii) an improved and definitive diagnosis and subsequent treatment.
Likelihood ratio of the proposed pathway (i.e. wrist MRI group) in the detection of scaphoid fracture compared to the current pathway (no further imaging group) | 3 months
  The overall likelihood ratio and diagnostic accuracy (sensitivity and specificity) of the MRI for the early identification of scaphoid fractures in the proposed pathway will be assessed against a 3-month conventional 4-view plain x-ray as the comparator.
Time (measured in days) taken to reach a definitive diagnosis and the first major treatment decision based on the MRI in comparison to the current pathway | 3 months
  The study will evaluate the time required to achieve a definitive diagnosis and deliver the subsequent appropriate treatment. It is considered that a definitive diagnosis is reached once there is agreement between the initial (at A&E/UCC) and/or the follow-up (at fracture clinic) imaging exams and the final 3-month plain x-ray.
Percentage of agreement between radiographers and radiologists in the diagnosis of suspected scaphoid fractures | 1 week
  The percentage of agreement between radiographers and radiologists in the diagnosis of suspected scaphoid fractures (i.e. rule in/rule out) using MRI datasets will also be assessed. This information will provide pivotal insight as to how the proposed clinical pathway can operationally be rolled out, as well as future areas of research.
Time off work or informal care needs (measured in days) due to the suspected scaphoid fracture. | 3 months
  The study aims to assess potential benefits from a broader societal perspective. For this purpose, time off work and informal care required due to the suspected scaphoid fracture will be recorded. The underlying hypothesis is that the use of MRI might reduce the amount of unnecessary plaster casts (i.e. in patients with no scaphoid fracture) and translate into a reduction in days off work and subsequent need for informal care.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Gidwani, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rua T, Vijayanathan S, Parkin D, Goh V, McCrone P, Gidwani S. Rationale and design of the SMaRT trial: A randomised, prospective, parallel, non-blinded, one-centre trial to evaluate the use of magnetic resonance imaging in acute setting in patients presenting with suspected scaphoid fracture. Clin Trials. 2018 Apr;15(2):120-129. doi: 10.1177/1740774517748320. Epub 2018 Jan 24. PMID 29366329